CLINICAL TRIAL: NCT04109820
Title: Effect of MitoQ on Platelet Function and Reactive Oxygen Species (ROS) Generation in Patients With Sickle Cell Anemia
Brief Title: Effect of MitoQ on Platelet Function and Reactive Oxygen Species Generation in Patients With Sickle Cell Anemia
Acronym: MitoQ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Ramasubramanian Kalpatthi, Assistant Professor, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY18120144
Record Dates: First submitted 2019-08-27; First posted 2019-09-30 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Sickle Cell Disease
Keywords: Basal platelet activation; MitoQ; mitochondrial ROS (Reactive Oxygen Species)
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — mitoquinone

STUDY DESIGN:
Intervention Model Description: Non randomized case control study design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sickle cell patients (Experimental): Sickle Cell subjects administered oral MitoQ (20mg once a day for 14 days)
  Interventions: Dietary Supplement: MitoQ
- Non Sickle cell Control subjects (Active Comparator): Normal control subjects administered oral MitoQ (20mg once a day for 14 days)
  Interventions: Dietary Supplement: MitoQ

INTERVENTIONS:
Dietary Supplement: MitoQ — Oral; 20mg once a day for 14 days

SUMMARY:
MitoQ is commercially available as a dietary supplement and it has been tested as a potential drug in other diseases, but it has never been tested in patients with sickle cell disease.

The goal of this research is to study if MitoQ, a molecule that works as an antioxidant by removing potentially damaging agents in a living organism, improves platelet function in patients with sickle cell disease (SCD).

DETAILED DESCRIPTION:
Antioxidant therapies targeted to specific enzymes or compartments may be beneficial in sickle cell anemia (SCA). MitoQ, the most extensively studied mitochondrial-targeted antioxidant, has been shown to be protective against ischemia/reperfusion injury in the heart, endothelial damage due to hypertension and ROS in animal models. MitoQ is commercially available as a dietary supplement to reduce overall oxidative stress and anti-ageing. However, MitoQ has not been tested either as a platelet antagonist or as an endothelial protectant in SCA patients. Investigators propose to conduct a small clinical trial of MitoQ in subjects with SCA to test the hypothesis that MitoQ scavenges platelet mtROS to prevent platelet activation and attenuate vascular dysfunction in SCA.

Investigators will test whether MitoQ decreases basal platelet activation in SCD patients and attenuates vascular dysfunction in subjects with SCA. Investigators will administer MitoQ orally to patients and healthy controls for 14 days. Investigators will obtain platelet count, hemolytic markers, platelet mtROS levels and activation markers, clinic BP measurements before and after MitoQ.

Adult male and female SCA subjects in steady state (n=10) and 5 healthy African-American volunteers will be recruited after obtaining informed consent.

ELIGIBILITY:
Inclusion Criteria:

Subjects

* African American
* Patients with sickle cell anemia
* 18 years old or older

Control

* African American healthy controls
* 18 years of age or older

Exclusion Criteria:

1. Pregnancy,
2. Known hypertension,
3. Hemodialysis and active obstructive sleep apnea requiring treatment.
4. Use of anti-platelet medication or have had transfusion in the 4 weeks prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Effect of MitoQ on platelet activation markers in subjects with SCA | Baseline to 14 days
  Change in the percentage of platelet activation markers in blood will be measured (p-selectin, activated GpIIb/IIIa expression, platelet mtROS [mitochondrial reactive oxygen species], platelet bioenergetics, mitochondrial Complex V activity)

SECONDARY OUTCOMES:
Effect of MitoQ on vascular dysfunction in subjects with SCA | Baseline to 14 days
  Changes in both systolic and diastolic blood pressure will be measured during the study period
Effect of MitoQ on hemolysis in subjects with SCA | Baseline to 14 days
  Changes in plasma free hemoglobin level (mg/dL) will be measured in blood.
Effect of MitoQ on hemolysis in subjects with SCA | Baseline to 14 days
  Changes in plasma adenosine diphosphate level (micromole/liter) will be measured in blood.
Effect of MitoQ on hemolysis in subjects with SCA | Baseline to 14 days
  Changes in serum lactate dehydrogenase level (units/L) will be measured in blood.
Treatment related severe adverse events (SAE) | Baseline to 14 days
  Overall incidence of treatment emergent severe adverse events (SAE)

CONTACTS AND LOCATIONS:
Overall Officials: Ramasubramanian Kalpatthi, MD, Principal Investigator — University of Pittsburgh
Locations (5):
- United States (5):
  - Magee Women's Hospital, Pittsburgh, Pennsylvania
  - UPMC Montefiore, Pittsburgh, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Hillman Cancer Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The investigators may share de-identified data with others who are doing similar types of research. All collected individual participant data (IPD), all IPD that underlie results in a publication will be shared.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available 6 months after the publication. July 2022.
Access Criteria: The IPD and any additional supporting information will be shared, with other investigators/collaborators when requested. The Principal Investigator will review the requests and will provide the instructions to the research site staff to share the IPD with other investigators.